CLINICAL TRIAL: NCT04947878
Title: Development and Validation of an Orthopedic Visit Prompt List
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, David Ring, MD, PhD Associate Dean for Comprehensive Care, Professor of Surgery and Psychiatry, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-0122
Record Dates: First submitted 2021-06-13; First posted 2021-07-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Musculoskeletal Diseases
Keywords: Orthopedics
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: All new, adult (18+ years old) patients seeing an orthopedic surgeon for a consultation will be invited to enroll. Randomization will be done through an Excel random number generator. The patients in the intervention group will review a prompt list before their visit. The research assistant will shadow the surgeon to count the amount of questions they ask during their visit. Patients in both groups will fill out a survey entailing demographics, the Decisional Conflict Scale, the JSPPE, the PAM score and a satisfaction scale at the end of the visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): will not review a prompt list before their visit.
- Prompt list (Experimental): The patients in the intervention group will review a prompt list before their visit.
  Interventions: Other: Prompt list

INTERVENTIONS:
Other: Prompt list — The patients in the intervention group will review a prompt list before their visit.
  Arms: Prompt list

SUMMARY:
Investigators are interested to see whether patients who received a visit question prompt list before the consultation ask more questions, feel more actively involved in their healthcare, and think of their surgeon as being more empathetic.

DETAILED DESCRIPTION:
Visiting a doctor with a musculoskeletal problem can be quite a daunting experience for patients. A visit question prompt list may help to empower patients and increase their role in active decision-making. Previous studies have shown that patient activation is correlated with a disability, pain intensity, and satisfaction with treatment. Perceived empathy is strongly associated with satisfaction among people with arm problems. A list that prompts patients to ask about things that matter to them, might improve their connection with the surgeon and their perceived empathy. The investigators are interested to see whether patients who received a visit question prompt list before the consultation ask more questions, feel more actively involved in their healthcare, and think of their surgeon as being more empathetic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+)
* Orthopedic visit

Exclusion Criteria:

* Patients who are illiterate.
* Patients who do not speak English.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | Baseline
  Questionnaire assessing decision conflict

SECONDARY OUTCOMES:
Jefferson Scale of Patient's Perceptions of Physician Empathy | Baseline
  Patient perceived of physician empathy as measured by the JSPPE
Patient Activation Measure-13 | Baseline
  Patient activation as measured by PAM-13
Satisfaction scale | Baseline
  Questionnaire measuring to what degree patients are satisfied with the care they received.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- UT health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No